CLINICAL TRIAL: NCT02028377
Title: Evaluation of the Novel Imaging Modality Simultaneous Positron Emission Tomography Magnetic Resonance Imaging (PET/MRI) in Patients With Pancreatic Adenocarcinoma
Brief Title: Evaluation of PET/MRI in Patients With Pancreatic Adenocarcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201212004
Record Dates: First submitted 2013-09-23; First posted 2014-01-07 (Estimated); Last update posted 2018-06-25 (Actual); Status verified 2018-06

CONDITIONS: Adenocarcinoma Pancreas
Keywords: Adenocarcinoma; imaging; PET; MRI
MeSH Terms: conditions — Adenocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Imaging (Experimental): PET/MRI
  Interventions: Procedure: PET/MRI

INTERVENTIONS:
Procedure: PET/MRI — PET/MRI

SUMMARY:
This study will use PET/MRI in patients with adenocarcinoma of the pancreas to identify hidden metastatic disease or identify patients with borderline or locally advanced disease.

DETAILED DESCRIPTION:
Patients will receive a PET/MRI scan within 6 weeks of their standard of care imaging. There is no maximum number of scans for research. The number of scans depends on each patient's treatment plan.

ELIGIBILITY:
Inclusion Criteria:

* Presence of suspicious lesion of the pancreas consistent with pancreatic adenocarcinoma. Cytological confirmation is not required.
* Patients preparing to receive therapy for pancreas cancer, including patients enrolled in NCT01413022
* Patient must be 18 years or older
* Patient must have a life expectancy of more than 6 months and performance status of 2 or less
* Patient must be able to understand and willing to sign an approved written informed consent document
* Women of childbearing potential and men must agree to use adequate contraception prior to study entry and for the length of the study
* Patients enrolled in the Clinical trials.gov# NCT01413022 trial must meet both studies eligibility criteria.

Exclusion Criteria:

* Patient must not have had prior resection for pancreatic adenocarcinoma.
* Patient must not have a history of other malignancy less than or equal to 5 years previous with the exception of basal cell or squamous cell carcinoma of the skin which were treated with local resection only or carcinoma in situ of the cervix
* Patient must not be unable to receive a PET-MRI scan due to renal function, allergy or other problem with receiving or tolerating an MRI scan, etc. All patients will fill out a standard MRI screening form.
* Patients must not have a blood glucose of greater than or equal to 200mg/dL at the time of PET-MRI or if a patient is diabetic and glucose is not controlled. At the discretion of the PI and the authorized user and with their approval prior to 2-[18]fluoro-2-deoxy-D-glucose (FDG) injection, patients with blood glucose ≥ 200 mg/dL may participate in the study.
* Patient must not be pregnant and/or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2017-08-22 (Actual); Study Completion 2017-08-22 (Actual)

PRIMARY OUTCOMES:
PET/MRI compared to conventional CT and MRI | Up to several months or longer. Patient will undergo research imaging with each standard of care scan they have.
  Primary outcome is to determine if the primary tumor and the margins of anatomical land marks from the PET/MRI imaging is more precise and gives a clearer picture of tumor location than standard care, CT or MRI. Both standard of care imaging and this new technology will be compared to the final pathologic analysis, measuring the true distance (in mm) between the primary tumor and margins. Data will be reported as mm.

SECONDARY OUTCOMES:
Resectability post neoadjuvant treatment | Several months or as deemed a surgical candidate by physician.
  The secondary outcome is to determine if PET/MRI imaging is better than standard of care imaging (CT or MRI) after patients have received chemotherapy and to determine if they are surgical candidates. The objective is to determine if the primary tumor and the margins of anatomical land marks from the PET/MRI imaging is more precise and gives a clearer picture of tumor location than standard care, CT or MRI. Both standard of care imaging and this new technology will be compared to the final pathologic analysis, measuring the true distance (in mm) between the primary tumor and margins. Data will be reported as mm.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan C. Fields, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington Unviversity School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Per, XII.1 and 2, Name and contact information will be kept for future research.